CLINICAL TRIAL: NCT06434506
Title: Prevalence and Risk Factors Associated With Wire Syndrome
Brief Title: Prevalence of the Wire Syndrome
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Odonto01
Record Dates: First submitted 2024-01-29; First posted 2024-05-30 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-01

CONDITIONS: Orthodontic Wires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NWS group: non-wire syndrome group
  Interventions: Other: no intervention
- WS group: wire syndrome group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention

SUMMARY:
The Wire Syndrome problem referred to dental displacements that can be described as aberrant, inaccurate, unexplained, or excessive on teeth still contained by an intact orthodontic wire, without detachment or fracture, leading to evolving dental and periodontal, aesthetic and/or functional consequences. The objective of this study was to define the prevalence of mandibular wire syndrome and the associated risk factors.

ELIGIBILITY:
Inclusion Criteria:-students in their 4th, 5th, and 6th year of dental studies at the Côte d'Azur University

- have undergone orthodontic treatment and are wearing a fixed mandibular retainer from canine to canine.

Exclusion Criteria:'- orthodontic treatment in progress

* absence/fracture of orthodontic fixed mandibular retainer
* wearing a removable mandibular retainer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: students in their 4th, 5th, and 6th year of dental studies at the Côte d'Azur University who have undergone orthodontic treatment and are wearing a fixed mandibular retainer from canine to canine
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of the Wire Syndrome | End : July 2023
  The prevalence of wire syndrome is the number of people affected by the wire syndrome at a given time in a given population. The prevalence rate is calculated by dividing this number of cases by the size of the exposed population. This study was design as a cross-sectional study conducted in the Orthodontics Unit of the Nice University Hospital from July 2022 to July 2023.

SECONDARY OUTCOMES:
Identify risk factors associated with wire syndrome - questionnaire | End : July 2023
  Questionnaire: 20 clinical questions without score
Identify risk factors associated with wire syndrome - clinical examination periodontium | End : July 2023
  Intraoral clinical examination:
  type of periodontium: thin and scalloped or flat and thick
Identify risk factors associated with wire syndrome - clinical examination - Angle | End : July 2023
  Intraoral clinical examinations:
  molar and canine relationships according to the Angle's classification class I, class II, Class III
Identify risk factors associated with wire syndrome - clinical examination: overbite / overjet | End : July 2023
  Intraoral clinical examinations:
  overbite and overjet in milimeters
Identify risk factors associated with wire syndrome - clinical examination / presence/absence clinical signs | End : July 2023
  Intraoral clinical examinations:
  presence/absence of an incisal guidance (YES / NO), presence/absence of parafunctions signs, (YES / NO)
Identify risk factors associated with wire syndrome - clinical examination / description clinical signs | End : July 2023
  Intraoral clinical examinations:
  clinical signs: observations : swallowing and tongue (no score / no mesure : only clinical observations)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Charavet, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No